CLINICAL TRIAL: NCT03047850
Title: Comparison of Delta Pulse Pressure and Delta Down Before and After Sternotomy
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, FCCP, Principal Investigator, Astes
Other Study IDs: DPPDD
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Hemodynamics
Keywords: Sternotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: All patients included in this study.
  Interventions: Diagnostic Test: Comparison of Delta Down and Delta Pulse Pressure

INTERVENTIONS:
Diagnostic Test: Comparison of Delta Down and Delta Pulse Pressure — Comparison of Delta Down and Delta Pulse Pressure Before and After Sternotomy.

SUMMARY:
Delta Pulse Pressure and Delta Down have been validated in surgery upon closed chest. This study aim to evaluate the influence of sternotomy on the value of Delta Pulse Pressure and Delta Down.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for open chest surgery.

Exclusion Criteria:

* Age < 18 years
* Patients with arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for open chest surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change of Delta Pulse Pressure Value | 10 minutes
  Change of Delta Pulse Pressure Value before and after sternotomy.
Change of Delta Down Value | 10 minutes
  Change of Delta Down before and after sternotomy.

CONTACTS AND LOCATIONS:
Overall Officials: Eric DEFLANDRE, MD, FCCP, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc of Bouge, Bouge, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No